CLINICAL TRIAL: NCT05355675
Title: The Association of Microbiota Composition With Chronic Graft Versus Host Disease
Brief Title: The Association of Microbiota Composition With cGVHD After Allo-HSCT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Principal Investigator, Yi Luo, Principal Investigator, First Affiliated Hospital of Zhejiang University
Other Study IDs: ZJU-HSCT-microbe
Record Dates: First submitted 2022-04-20; First posted 2022-05-02 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Hematopoietic Stem Cell Transplantation; Hematologic Malignancy; Chronic Graft-versus-host-disease; Complication
Keywords: hematopoietic stem cell transplantation; microbiota; metabolomics; chronic graft versus host disease
MeSH Terms: conditions — Hematologic Neoplasms; Bronchiolitis Obliterans Syndrome | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — This blood will be used for plasma banking for further analysis, including miR and chemokine detection. Stool will be used for microbiome studies - isolation of total DNA/RNA and 16S rRNA gene sequencing for bacterial taxonomic classification. Furthermore, metagenomic sequencing and subsequent taxonomic and functional classification of microbial genes will be used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- observational group: Patients with hematologic malignancies following allogeneic hematopoietic stem cell transplantation treatment
  Interventions: Other: blood sample; Other: stool sample
- control group: health control group: healthy volunteers
  Interventions: Other: blood sample; Other: stool sample

INTERVENTIONS:
Other: blood sample — collecting 15ml peripheral blood samples at -7 days before transplantation and+28 days, +100 days, +1 years, +2 years after transplantation
Other: stool sample — collecting 50mg fresh stool samples at -7 days before transplantation and+28 days, +100 days, +1 years, +2 years after transplantation

SUMMARY:
Previous studies had found that the microbe in intestinal after allogeneic hematopoietic cell transplantation(allo-HSCT) were closely associated with overall survival and post-transplantation complications, especially graft versus host disease (GVHD).Due to the limited data on the association of microbiota composition with chronic GVHD(cGVHD) after allogeneic hematopoietic stem cell transplantation, the relationship between microbiota composition and post-transplantation complications, especially cGVHD, needs to be further evaluated.Detailed studies of the microbiome and host immune system will lead to the discovery of microbiome markers for early identification of patients at high risk for cGVHD. This may regulate patients' gut microbiota in an individualized manner to achieve optimal treatment outcomes while avoiding severe post-transplant cGVHD. We will operate a prospective, multicenter, nonrandomized, observational study. Patients will be asked to provide blood and stool samples during allo-HSCT.

DETAILED DESCRIPTION:
Previous studies had found that the microbe in intestinal after allogeneic hematopoietic cell transplantation(allo-HSCT) were closely associated with overall survival and post-transplantation complications, especially graft versus host disease (GVHD).Due to the limited data on the association of microbiota composition with chronic GVHD(cGVHD) after allogeneic hematopoietic stem cell transplantation, the relationship between microbiota composition and post-transplantation complications, especially cGVHD, needs to be further evaluated.Detailed studies of the microbiome and host immune system will lead to the discovery of microbiome markers for early identification of patients at high risk for cGVHD. This may regulate patients' gut microbiota in an individualized manner to achieve optimal treatment outcomes while avoiding severe post-transplant cGVHD. We will operate a prospective, multicenter, nonrandomized, observational study. Patients will be asked to provide blood and stool samples during allo-HSCT. This blood will be used for plasma banking for further analysis, including miR, chemokine and metabonomics detection. Stool will be used for microbiome studies - isolation of total DNA/RNA and 16S rRNA gene sequencing for bacterial taxonomic classification. Furthermore, metagenomic sequencing and subsequent taxonomic and functional classification of microbial genes will be used.

ELIGIBILITY:
Inclusion Criteria:

1. aged between 18 years and 65 years
2. patients planned to be treated by allogeneic hematopoietic cell transplantation
3. signed written informed consent

Exclusion Criteria:

patients not-matching inclusion criteria

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with hematologic malignancies planned to be treated by allogeneic hematopoietic cell transplantation
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Microbial changes in stool as measured by 16S rRNA gene sequencing in hematological cancer patients before, at time and after hematopoietic cell transplantation | 100 days
  Microbial changes of stool will be assessed before, at time and after hematopoietic cell transplantation

SECONDARY OUTCOMES:
To correlate microbial changes in stool as measured by 16S rRNA gene sequencing with the post-transplant complications in allogeneic transplant settings (cGVHD, overall survival, non-relapse mortality, replase, infectious complications) | 100 days
  To assess microbial changes with toxicity of therapy
To correlate microbial changes in stool as measured by 16S rRNA gene sequencing with the patients reported outcomes | 100 days
  To correlate microbial changes with the quality of life which measured by Short Form 36 (SF-36) and and Functional Assessment of Chronic Illness Therapy with BMT subscale (FACT-BMT)
To correlate microbial changes in stool as measured by 16S rRNA gene sequencing with the patients nutrition status | 100 days
  To correlate microbial changes with the patients nutrition. Clinical and biological nutritional assessments included anthropometric measurements, serum nutritional proteins, body composition assessed by bioelectrical impedance, and upper-limb muscle strength (MS) measured by dynamometry.

CONTACTS AND LOCATIONS:
Overall Officials: Yi Luo, M.D., Principal Investigator — First Affilaated Hospital of Medical School of Zhejiang University
Locations (9):
- China (9):
  - The first Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - First Affiliated Hospital of Zhejiang Chinese Medicine University, Hangzhou, Zhejiang
  - Second Affiliated Hospital of Zhejiang University, School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, College of Medicine, Zhejiang University, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - Jinhua Hospital of Zhejiang University, Jinhua
  - Ningbo Hospital of Zhejiang University, Ningbo
  - The Affiliated People's Hospital of Ningbo University, Ningbo
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou

IPD SHARING:
Plan to Share IPD: No